CLINICAL TRIAL: NCT05094765
Title: Evaluating Safety and Efficacy of GI-XBI-302 in Patients With Glucocorticoid-refractory Acute Graft vs. Host Disease After Allogeneic Stem Cell Transplantation
Brief Title: Fecal Microbiota Transplant (FMT) Capsule for Improving the Efficacy of GI-aGVHD
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Xbiome Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XCT4843002
Record Dates: First submitted 2021-09-29; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-09

CONDITIONS: GVHD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT (Experimental): 60 capsules per day for 2 day
  Interventions: Biological: FMT

INTERVENTIONS:
Biological: FMT — Fecal Microbiota Transplantation

SUMMARY:
This study aims to determine whether the fecal microbiota transplant (FMT) capsule improves the response rate of GI-aGVHD in patients with glucocorticoid-refractory acute graft vs. host disease after allogeneic stem cell transplantation

ELIGIBILITY:
Inclusion Criteria:

* 1. GVHD within 100 days after allogeneic hematopoietic stem cell transplantation (allo HSCT);

  2. Age 18 - 65 years old, regardless of gender;

  3. Patients with grade 3 or 4 gastrointestinal involvement (aGVHD) according to the International Alliance (Magic) classification standard;

  4. Patients with glucocorticoid resistant GI aGVHD are diagnosed. According to the expert consensus of Chinese allogeneic hematopoietic stem cell transplantation for the treatment of hematological diseases (III) - acute graft-versus-host disease (2020 Edition), the definition of glucocorticoid resistant acute GVHD is Thomas' hematopoietic cell transplantation: stem cell transplantation (5th Edition) Glucocorticoid resistance was defined as PD at 3 days, NR at 7 days or Cr not reached at 14 days after first-line treatment.

  5. ECoG 3 points or less;

  6. Stop prophylactic antibiotics at least 12 hours before FMT treatment;

  7. Be able and willing to sign informed consent;

  8. Patients who are capable of swallowing capsules and can complete the study;

Exclusion Criteria:

* 1. There are active but uncontrolled infections, except GVHD complicated with infectious diarrhea;

  2. Gastrointestinal perforation, active gastrointestinal bleeding, small intestinal obstruction, toxic megacolon or other serious gastrointestinal diseases not caused by GVHD;

  3. Have a history of severe allergic reaction; Or known to be allergic to any ingredient of intestinal bacteria capsule xbi-302;

  4. Any serious disease that can increase the risk of patients participating in the study;

  5. Female subjects with positive pregnancy test and lactation, or female subjects of childbearing age who refuse to take contraceptive measures during the study;

  6. According to the judgment of the researcher, the patients with high dynamic diarrhea can not stay in the intestine for enough time to dissolve the capsule.

  7. HIV, HBV, HCV and syphilis are positive;

  8. After colectomy;

  9. Participate in other intervention clinical studies within 4 weeks before the screening period;

  10. The expected survival time is less than 12 weeks;

  11. The basic body function test is inferior to the following standards: total neutrophils (neu) < 0.5 (x109 / L), platelet count (PLT) < 30 (x109 / L), serum creatinine (CR) > 1.5 times the maximum normal value (ULN), albumin (ALB) < 25g / L;

  12. There is any situation that the researcher thinks is not suitable for inclusion (any history of medical history, treatment history or abnormal test data that may confuse the results of this study, interfere with the subject's whole participation in the study, or harm the interests of the subject).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-03-02 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
ORR | Day 28
  assessed by Overall Response Rate (ORR) at Day 28
AE | Day 28
  assessed all related a grade 3 or above adverse event (AE) at Day 28

SECONDARY OUTCOMES:
AE | up to 25 weeks
  assessed all related adverse event (AE)
Shannon index | up to 25 weeks
  changes of Shannon index
colonization bacteria analysis | up to 25 weeks
  the number and relative abundance of bacteria that originally existed only in the capsule but could still be detected in the stool samples of subjects
PFS | up to 25 weeks
  Kaplan-Meier Curve

OTHER OUTCOMES:
Metabonomics | up to 25 weeks
  The changes of calprotectin, Is, SCFA and bile acid were compared
biomarkers | up to 25 weeks
  The changes of IL-6、IL-8、sTNFR1、sST2、Reg3a、Elafin were compared
Immunohistochemistry | up to 25 weeks
  The phenotypes and subsets of CD4 and CD8 positive T cells, B cells, NK cells and monocytes were compared
Proportion of patients | up to 25 weeks
  Proportion of patients with hormone dosage ≤ 20mg / day equivalent to equivalent converted dose of prednisolone
The proportion of patients | up to 25 weeks
  who stopped antibiotics was compared.
Percentage of patients | up to 25 weeks
  Percentage of patients who died due to GVHD

IPD SHARING:
Plan to Share IPD: Undecided